CLINICAL TRIAL: NCT03085797
Title: A Randomised, Double-blind, Parallel Group PhIII Study to Assess the Clinical Efficacy and Safety of 100 mg SC Mepolizumab as an Add on to Maintenance Treatment in Adults With Severe Bilateral Nasal Polyps - SYNAPSE (StudY in NAsal Polyps Patients to Assess the Safety and Efficacy of Mepolizumab)
Brief Title: Effect of Mepolizumab in Severe Bilateral Nasal Polyps
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: CRF Health (Industry); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 205687; 2016-004255-70 (EudraCT Number)
Record Dates: First submitted 2017-03-15; First posted 2017-03-21 (Actual); Results first posted 2020-12-17 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-08

CONDITIONS: Nasal Polyps
Keywords: SB240563; Nasal Polyps; Mepolizumab; Phase 3; Parallel group; Efficacy
MeSH Terms: conditions — Nasal Polyps | interventions — mepolizumab; Mometasone Furoate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Mepolizumab 100 mg SC + MF (Experimental): Participants will receive total thirteen doses of 100 mg SC of mepolizumab in thigh, abdomen or upper arm every 4 weeks for 52 weeks on top of SoC which includes daily nasal spray of mometasone furoate.
  Interventions: Drug: Mepolizumab; Drug: Mometasone furoate
- Placebo SC + MF (Placebo Comparator): Participants will receive total thirteen doses of SC matching placebo in thigh, abdomen or upper arm every 4 weeks for 52 weeks on top of SoC which includes daily nasal spray of mometasone furoate.
  Interventions: Drug: Placebo; Drug: Mometasone furoate

INTERVENTIONS:
Drug: Mepolizumab — Mepolizumab injection 100 mg/millilitre (mL) is a clear to opalescent, colorless to pale yellow to pale brown sterile solution for SC injection in a single-use, safety syringe.
  Arms: Mepolizumab 100 mg SC + MF
Drug: Placebo — Placebo is a clear to opalescent, colorless sterile solution for SC injection in a single-use, safety syringe.
  Arms: Placebo SC + MF
Drug: Mometasone furoate — All participants will receive mometasone furoate usually 400 micrograms (mcg), 2 actuations (50 mcg/actuation) in each nostril twice daily. Intolerant participants will use 200g (2 actuations [50 g/actuation] in each nostril once daily).

SUMMARY:
Nasal polyps (NP) has long been known as chronic inflammatory disease of the nasal mucosa. This disease is characterized by the presence of polyps in the upper nasal cavity, originating from within the ostiomeatal complex. The presence of polyps can cause long-term symptoms such as prominent nasal obstruction, post-nasal drip, loss of smell, and discharge.

Mepolizumab (SB240563) is an Immunoglobulin G 1 [IgG1], kappa humanized monoclonal antibody (mAB) that blocks human interleukin-5 (hIL-5) from binding to the interleukin-5 (IL-5) receptor complex expressed on the eosinophil cell surface and thus inhibits signaling. Neutralization of IL-5 with mepolizumab has been shown to reduce blood, sputum and tissue eosinophils and hence is assumed to be a treatment option in a number of eosinophilic diseases including NP.

The aim of this randomized, double-blind, parallel group, phase 3 (PhIII) study is to assess the clinical efficacy and safety of 100 milligram (mg) subcutaneous (SC) mepolizumab as an add on to maintenance treatment in adults with severe bilateral NP. The study will include a 4-week run in period followed by randomization to a 52-week treatment period. Participants will receive mepolizumab 100 mg or placebo SC by the investigator or delegate via a pre-filled safety syringe every 4 weeks for 52 weeks. Throughout the entire study period (run in + treatment period + follow up), participants will receive a standard of care (SoC) for NP which consists of daily mometasone furorate (MF) nasal spray, and if required, saline nasal douching, occasional short courses of high dose oral corticosteroids (OCS) and/or antibiotics. The treatment period will consist of thirteen, 4-weekly doses of mepolizumab or placebo. In addition, up to the first 200 randomized participants will be followed up every other month for up to a further 6 months after the Visit 15 (7 months post last dose) in order to assess maintenance of response and to validate a physiological model derived from the previous Phase 2 study. Approximately 400 participants will be randomized (200 participants per treatment arm) in to the study. Total duration of the study will be 76 weeks for first 200 randomized participants and 52 weeks for remainder of participants who are not participating in the 6 months no treatment follow up.

ELIGIBILITY:
Inclusion Criteria

* 18 years of age and older inclusive, at the time of signing the informed consent.
* Body weight greater or equal to 40 kilogram (kg).
* Male or female participants (with appropriate contraceptive methods) to be eligible for entry into the study. To be eligible for entry into the study, woman of childbearing potential (WOCBP) must commit to consistent and correct use of an acceptable method of birth control from the time of consent, for the duration of the trial, and for 105 days after last study drug administration.
* Participants who have had at least one previous surgery in the previous 10 years for the removal of NP. NP Surgery is defined as any procedure involving instruments with resulting incision (cutting open) and removal of polyp tissue from the nasal cavity (polypectomy). For the purpose of inclusion into this study, any procedure involving instrumentation in the nasal cavity resulting in dilatation of the nasal passage such as balloon sinuplasty, insertion of coated stents or direct injection of steroids or other medication without any removal of NP tissue is not accepted.
* Participants with bilateral NP as diagnosed by endoscopy or computed tomography (CT) scan.
* Presence of at least two of the following symptoms one of which should be either nasal blockage/obstruction/congestion or nasal discharge (anterior/posterior nasal drip) and either nasal discharge (anterior/posterior nasal drip); facial pain/pressure; reduction or loss of smell for at least 12 weeks prior to screening.
* Participants with severe NP symptoms defined as an obstruction VAS symptom score of >5.
* Severity consistent with a need for surgery as described by:

  1. Participants with an overall VAS symptom score >7,
  2. Participants with an endoscopic bilateral NP score of at least 5 out of a maximum score of 8 (with a minimum score of 2 in each nasal cavity).
* Treatment with intranasal corticosteroids (INCS) for at least 8 weeks prior to screening.
* Capable of giving signed informed consent Exclusion Criteria
* As a result of medical interview, physical examination, or screening investigation, the physician responsible considers the participant unfit for the study.
* Cystic fibrosis
* Eosinophilic granulomatosis with polyangiitis (also known as churg strauss syndrome), young's, kartagener's or dyskinetic ciliary syndromes.
* Antrochoanal polyps
* Nasal septal deviation occluding one nostril
* Acute sinusitis or upper respiratory track infection (URTI) at screening or in 2 weeks prior to screening
* Ongoing rhinitis medicamentosa (rebound or chemical induced rhinitis)
* Participants who have had an asthma exacerbation requiring admission to hospital within 4 weeks of Screening.
* Participants who have undergone any intranasal and/or sinus surgery (for example polypectomy, balloon dilatation or nasal stent insertion) within 6 months prior Visit 1.
* Participants where NP surgery is contraindicated in the opinion of the Investigator.
* Participants with a known medical history of human immunodeficiency virus (HIV) infection.
* Participants with a known, pre-existing parasitic infestation within 6 months prior to Visit 1.
* Participants who are currently receiving, or have received within 3 months (or 5 half lives - whatever is the longest) prior to first mepolizumab dose, chemotherapy, radiotherapy or investigational medications/therapies.
* Participants with a history of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK medical monitor, contraindicates their participation. Aspirin-sensitive participants are acceptable.
* Participants with a history of allergic reaction to anti-IL-5 or other monoclonal antibody therapy.
* Participants on a waiting list for NP surgery while at screening
* Participants that have taken part in previous mepolizumab, reslizumab, dupilumab or benralizumab studies.
* Use of systemic corticosteroids (including oral corticosteroids) or corticosteroid nasal solution (intranasal corticosteroid is accepted) within 4 weeks prior to Screening or planned use of such medications during the double-blind period.
* INCS dose changes within 1 month prior to screening.
* Treatments with biological or immunosuppressive treatment (other than omalizumab) treatment within 5 terminal phase half lives of Visit 1.
* Omalizumab treatment in the 130 days prior to Visit 1.
* Commencement of leukotriene antagonist treatment less than 30 days prior to Visit 1.
* Allergen immunotherapy within the previous 3 months.
* Women who are pregnant or lactating or are planning on becoming pregnant during the study.
* Participants who currently smoke or have smoked in the last 6 months.
* Any participant who is considered unlikely to survive the duration of the study period or has any rapidly progressing disease or immediate life-threatening illness (e.g. cancer). In addition, any participant who has any other condition (e.g. neurological condition) that is likely to affect respiratory function should not be included in the study.
* Participants who have known, pre-existing, clinically significant endocrine, autoimmune, cardiovascular, metabolic, neurological, renal, gastrointestinal, hepatic, hematological or any other system abnormalities that are uncontrolled with standard treatment.
* Immunocompromized, other than that explained by the use of corticosteroids taken as therapy.
* A current malignancy or previous history of cancer in remission for less than 12 months prior to Screening. Participants with successfully treated basal cell carcinoma, squamous cell carcinoma of the skin, or cervical carcinoma in situ, with no evidence of recurrence may participate in the study.
* Current active liver or biliary disease (with the exception of gilbert's syndrome or asymptomatic gallstones or otherwise stable chronic liver disease per investigator assessment).
* Corrected QT interval (QTc) >450 milliseconds (msec) or QTc >480 msec in participants with bundle branch block at visit 1.
* A known or suspected history of alcohol or drug abuse within 2 years prior to Screening (Visit 1) that in the opinion of the investigator would prevent the participant from completing the study procedures.
* An investigator, sub-investigator, study coordinator, employee of a participating investigator or study site, or immediate family member of the aforementioned that is involved in this study.
* In the opinion of the investigator, any participant who is unable to read and/or would not be able to complete a questionnaire.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 414 (Actual)
Dates: Start 2017-05-25 (Actual); Primary Completion 2019-12-11 (Actual); Study Completion 2019-12-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (84):
- United States (34):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Riverside, California
  - GSK Investigational Site, Roseville, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Colorado Springs, Colorado
  - GSK Investigational Site, Lake Mary, Florida
  - GSK Investigational Site, Boise, Idaho
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Des Moines, Iowa
  - GSK Investigational Site, West Des Moines, Iowa
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Marrero, Louisiana
  - GSK Investigational Site, White Marsh, Maryland
  - GSK Investigational Site, Columbia, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Piscataway, New Jersey
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Matthews, North Carolina
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Medford, Oregon
  - GSK Investigational Site, Bethlehem, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Orangeburg, South Carolina
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, McKinney, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, North Logan, Utah
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, Lynchburg, Virginia
  - GSK Investigational Site, Norfolk, Virginia
  - GSK Investigational Site, Richmond, Virginia
- Argentina (8):
  - GSK Investigational Site, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - GSK Investigational Site, Florida, Buenos Aires
  - GSK Investigational Site, La Plata, Buenos Aires
  - GSK Investigational Site, Mar del Plata, Buenos Aires
  - GSK Investigational Site, Rosario, Santa Fe Province
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Mendoza
  - GSK Investigational Site, San Miguel de Tucumán
- Australia (5):
  - GSK Investigational Site, Darlinghurst, New South Wales
  - GSK Investigational Site, Westmead, New South Wales
  - GSK Investigational Site, Clayton, Victoria
  - GSK Investigational Site, Melbourne, Victoria
  - GSK Investigational Site, Murdoch, Western Australia
- Canada (7):
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Hamilton, Ontario
  - GSK Investigational Site, London, Ontario
  - GSK Investigational Site, Ottawa, Ontario
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Saskatoon, Saskatchewan
  - GSK Investigational Site, Québec
- Germany (8):
  - GSK Investigational Site, Tübingen, Baden-Wurttemberg
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Wiesbaden, Hesse
  - GSK Investigational Site, Düsseldorf, North Rhine-Westphalia
  - GSK Investigational Site, Münster, North Rhine-Westphalia
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Lübeck, Schleswig-Holstein
  - GSK Investigational Site, Berlin
- GSK Investigational Site, Amsterdam, Netherlands
- Romania (4):
  - GSK Investigational Site, Brasov
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Cluj-Napoca
  - GSK Investigational Site, Târgu Mureş
- Russia (4):
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Saint-Peterburgh
  - GSK Investigational Site, Yaroslavl
- South Korea (3):
  - GSK Investigational Site, Incheon
  - GSK Investigational Site, Seongnam-si Gyeonggi-do
  - GSK Investigational Site, Seoul
- Sweden (4):
  - GSK Investigational Site, Gothenburg
  - GSK Investigational Site, Helsingborg
  - GSK Investigational Site, Lund
  - GSK Investigational Site, Stockholm
- United Kingdom (6):
  - GSK Investigational Site, Darlington, Durham
  - GSK Investigational Site, Liverpool, Merseyside
  - GSK Investigational Site, London
  - GSK Investigational Site, Manchester
  - GSK Investigational Site, Newcastle upon Tyne
  - GSK Investigational Site, Rotherham

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study is available via the Clinical Study Data Request site
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (copy the URL below to your browser)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=20845

REFERENCES:
- [Background] Han JK, Bachert C, Fokkens W, Desrosiers M, Wagenmann M, Lee SE, Smith SG, Martin N, Mayer B, Yancey SW, Sousa AR, Chan R, Hopkins C; SYNAPSE study investigators. Mepolizumab for chronic rhinosinusitis with nasal polyps (SYNAPSE): a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet Respir Med. 2021 Oct;9(10):1141-1153. doi: 10.1016/S2213-2600(21)00097-7. Epub 2021 Apr 16. PMID 33872587
- [Derived] Chupp G, Alobid I, Lugogo NL, Kariyawasam HH, Bourdin A, Chaker AM, Smith SG, Sousa AR, Mayer B, Chan RH, Matucci A. Mepolizumab Reduces Systemic Corticosteroid Use in Chronic Rhinosinusitis With Nasal Polyps. J Allergy Clin Immunol Pract. 2023 Nov;11(11):3504-3512.e2. doi: 10.1016/j.jaip.2023.08.015. Epub 2023 Aug 14. PMID 37586475
- [Derived] Fokkens W, Trigg A, Lee SE, Chan RH, Diamant Z, Hopkins C, Howarth P, Lund V, Mayer B, Sousa AR, Yancey S, Tabberer M; SYNAPSE study group. Mepolizumab improvements in health-related quality of life and disease symptoms in a patient population with very severe chronic rhinosinusitis with nasal polyps: psychometric and efficacy analyses from the SYNAPSE study. J Patient Rep Outcomes. 2023 Jan 20;7(1):4. doi: 10.1186/s41687-023-00543-5. PMID 36662344
- [Derived] Fokkens WJ, Mullol J, Kennedy D, Philpott C, Seccia V, Kern RC, Coste A, Sousa AR, Howarth PH, Benson VS, Mayer B, Yancey SW, Chan R, Gane SB. Mepolizumab for chronic rhinosinusitis with nasal polyps (SYNAPSE): In-depth sinus surgery analysis. Allergy. 2023 Mar;78(3):812-821. doi: 10.1111/all.15434. Epub 2022 Jul 27. PMID 35822924
- [Derived] Bachert C, Sousa AR, Han JK, Schlosser RJ, Sowerby LJ, Hopkins C, Maspero JF, Smith SG, Kante O, Karidi-Andrioti DE, Mayer B, Chan RH, Yancey SW, Chaker AM. Mepolizumab for chronic rhinosinusitis with nasal polyps: Treatment efficacy by comorbidity and blood eosinophil count. J Allergy Clin Immunol. 2022 May;149(5):1711-1721.e6. doi: 10.1016/j.jaci.2021.10.040. Epub 2022 Jan 7. PMID 35007624
- [Derived] Chong LY, Piromchai P, Sharp S, Snidvongs K, Webster KE, Philpott C, Hopkins C, Burton MJ. Biologics for chronic rhinosinusitis. Cochrane Database Syst Rev. 2021 Mar 12;3(3):CD013513. doi: 10.1002/14651858.CD013513.pub3. PMID 33710614
- [Derived] Keene ON. Strategies for composite estimands in confirmatory clinical trials: Examples from trials in nasal polyps and steroid reduction. Pharm Stat. 2019 Jan;18(1):78-84. doi: 10.1002/pst.1909. Epub 2018 Oct 29. PMID 30370691

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants (par.) were enrolled across 11 countries (Germany, Netherlands, Romania, Sweden, United Kingdom, United States, Argentina, Australia, Canada, Republic of Korea and Russian Federation).
Pre-assignment Details: A total of 414 participants were enrolled and randomized in the study, of which only 407 participants received study treatment and were included in the Intent-to-Treat Population (defined as all randomized participants who took at least 1 dose of study treatment). Seven participants did not receive study treatment as they were randomized in error.
Groups:
- Placebo: Participants were randomized to receive up to 13 subcutaneous (SC) doses of mepolizumab matching placebo every 4 weeks to Week 52 (Wk 52) on top of standard of care (SoC) for nasal polyps (NP) which included daily mometasone furorate nasal spray. By design, some randomized participants were eligible to enter a further 6-month no-treatment follow-up period to assess maintenance of response after cessation of treatment.
- Mepolizumab 100 mg SC: Participants were randomized to receive up to 13 SC doses of mepolizumab 100 milligrams per milliliter (mg/mL) every 4 weeks to Week 52 on top of SoC for nasal polyps which included daily mometasone furorate nasal spray. By design, some randomized participants were eligible to enter a further 6-month no-treatment follow-up period to assess maintenance of response after cessation of treatment.
Period: Treatment Period (TP) (52 Weeks)
Arm/Group | Placebo | Mepolizumab 100 mg SC
Started (Data presented for ITT Population) | 201 | 206
Completed Investigational Product (IP) | 167 | 183
Not Completed IP | 34 | 23
Withdrew IP Due to: Adverse Event | 4 | 4
Withdrew IP Due to: Lack of Efficacy | 11 | 5
Withdrew IP Due to: Protocol Deviation | 1 | 0
Withdrew IP Due to: Stopping Criteria | 1 | 1
Withdrew IP Due to: Physician Decision | 2 | 1
Withdrew IP Due to: Withdrawal by Par. | 15 | 12
Completed | 184 | 189
Not Completed | 17 | 17
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 16 | 17
Period: No-treatment Follow-up Period (6 Months)
Arm/Group | Placebo | Mepolizumab 100 mg SC
Started | 65 (Only 65 Par. continued in FU to check maintenance of response after stopping treatment per protocol) | 69 (Only 69 Par. continued in FU to check maintenance of response after stopping treatment per protocol)
Completed | 65 | 68
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Mepolizumab 100 mg SC | Total
Number analyzed (Participants) | 201 | 206 | 407
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.9 (12.46) | 48.6 (13.55) | 48.8 (13.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 67 | 143
  Male | 125 | 139 | 264
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian-Central/South Asian Heritage (H.) | 1 | 2 | 3
  Race: Asian-Japanese H./East Asian H./SouthEast Asian H. | 8 | 7 | 15
  Race: Black or African American (AA) | 4 | 5 | 9
  Race: White | 187 | 192 | 379
  Race: AA/African H. and American Indian or Alaska Native | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Total Endoscopic Nasal Polyps Score at Week 52
Description: Independent reviewers, blinded to treatment, reviewed image recordings of nasal endoscopies to determine total endoscopic NP score based on NP size. The right and left nostrils were scored from 0 to 4 (0 = No polyps; 1 = Small polyps in the middle meatus not reaching below the inferior border of the middle concha; 2 = Polyps reaching below the lower border of the middle turbinate; 3 = Large polyps reaching the lower border of the inferior turbinate or polyps medial to the middle concha; and 4 = Large polyps causing complete obstruction/congestion of the inferior meatus). The total score is the sum of the right and left nostril scores and ranges from 0 to 8, higher scores indicate greater disease severity. Data up to Week 52, including from participants who remained in the study after early discontinuation from IP, were included in analysis. Baseline was defined as Day 1 value. Change from Baseline = Post-baseline value minus Baseline value.
Time Frame: Baseline (Day 1) and Week 52
Population: ITT Population which included all randomized participants who took at least 1 dose of study treatment.
Measure: Median (Full Range); unit: Scores on a scale
Arm/Group | Placebo | Mepolizumab 100 mg SC
Number analyzed (Participants) | 201 | 206
Scores on a scale | 0.0 [-5 to 3] | -1.0 [-6 to 3]
Statistical Analysis 1: Comparison: Placebo vs Mepolizumab 100 mg SC; Test type: Superiority; p < 0.001, Wilcoxon rank-sum test — p-Value was based on Wilcoxon rank-sum test; Difference in Medians = -0.73, 95% CI 2-sided [-1.11 to -0.34] — Quantile regression with covariates: treatment,region,Baseline score,Baseline eosinophilcount(BEC). Par. with nasal surgery prior to Wk52/withdrew early with no nasal surgery assigned their worst observed score prior to nasal surgery/study withdrawal

2. Primary Outcome: Change From Baseline in Nasal Obstruction Visual Analog Scale (VAS) Score During the 4 Weeks Prior to Week 52
Description: Participants rated individual (nasal obstruction, nasal discharge, mucus in the throat, loss of smell, facial pain) and overall symptoms on a visual analog scale (VAS) using an electronic diary (eDiary). Captured scores ranged between 0 (none) and 100 (as bad as you can imagine), final scores derived from the electronically captured scores by dividing by 10. The final nasal obstruction VAS score ranged between 0 and 10, with higher scores indicating greater disease severity. Data up to Week 52, including from participants who remained in the study after early discontinuation from IP, were included in analysis. The average of daily scores in 4-weekly intervals were calculated and data is presented for Weeks 49-52. Baseline was defined as the average score from the 7 days of eDiary data collected prior to Day 1. Change from Baseline = Post-baseline value minus Baseline value.
Time Frame: Baseline and Weeks 49 to 52
Population: ITT Population
Measure: Median (Full Range); unit: Scores on a scale
Arm/Group | Placebo | Mepolizumab 100 mg SC
Number analyzed (Participants) | 201 | 206
Scores on a scale | -0.82 [-9.23 to 2.58] | -4.41 [-9.90 to 1.54]
Statistical Analysis 1: Comparison: Placebo vs Mepolizumab 100 mg SC; Test type: Superiority; p < 0.001, Wilcoxon rank-sum test — p-Value was based on Wilcoxon rank-sum test; Difference in Medians = -3.14, 95% CI 2-sided [-4.09 to -2.18] — Quantile regression with covariates: treatment, region, Baseline score, Baseline BEC. Par. with nasal surgery prior to Wks 49-52/withdrew early with no nasal surgery assigned their worst observed 4-wk mean prior to nasal surgery/study withdrawal

3. Secondary Outcome: Percentage of Participants With Nasal Surgery Over Time
Description: The percentage of participants with nasal surgery over time (by Weeks 8, 16, 24, 32, 40, 48 and 52) was derived from Kaplan-Meier time-to-event analyses for the event 'first nasal surgery'. Nasal surgery was defined as any procedure involving instruments resulting in incision and removal of tissue (polypectomy) in the nasal cavity. Time to first nasal surgery was defined as (Date of first nasal surgery - Date of first dose of study treatment) + 1. Percentage of participants with nasal surgery over time (by Weeks 8, 16, 24, 32, 40, 48 and 52) and corresponding 95% CI have been presented, calculated using the Kaplan-Meier method. Analysis included surgeries occurring up to Week 52, reported on-treatment and those reported after early discontinuation from IP by participants who remained in the study.
Time Frame: Weeks 8, 16, 24, 32, 40, 48 and 52
Population: ITT Population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | Mepolizumab 100 mg SC
Number analyzed (Participants) | 201 | 206
Percentage of participants
  Week 8 | 1.0 [0.3 to 3.9] | 0.5 [0.1 to 3.4]
  Week 16 | 3.5 [1.7 to 7.2] | 1.0 [0.2 to 3.8]
  Week 24 | 9.1 [5.8 to 14.0] | 4.0 [2.0 to 7.8]
  Week 32 | 14.2 [10.0 to 19.9] | 6.0 [3.5 to 10.4]
  Week 40 | 18.9 [14.0 to 25.1] | 7.6 [4.6 to 12.3]
  Week 48 | 22.0 [16.8 to 28.5] | 9.2 [5.9 to 14.2]
  Week 52 | 23.6 [18.3 to 30.3] | 9.2 [5.9 to 14.2]
Statistical Analysis 1: Comparison: Placebo vs Mepolizumab 100 mg SC; Test type: Superiority; p = 0.003, Cox Proportional Hazards Model — p-Value was based on Cox Proportional Hazards Model; Hazard Ratio (Mepolizumab/Placebo) = 0.43, 95% CI 2-sided [0.25 to 0.76] — Analysis using a Cox Proportional Hazards Model with covariates of treatment, geographic region, Baseline total endoscopic score (centrally read), Baseline nasal obstruction VAS, Baseline BEC, number of previous surgeries (1, 2, >2 as ordinal)

4. Secondary Outcome: Change From Baseline in Overall VAS Score During the 4 Weeks Prior to Week 52
Description: Participants rated individual (nasal obstruction, nasal discharge, mucus in the throat, loss of smell, facial pain) and overall symptoms on a visual analog scale using an eDiary. Captured scores ranged between 0 (none) and 100 (as bad as you can imagine), final scores derived from the electronically captured scores by dividing by 10. The final overall VAS score ranged between 0 and 10, with higher scores indicating greater disease severity. Data up to Week 52, including from participants who remained in the study after early discontinuation from IP, were included in analysis. The average of daily scores in 4-weekly intervals were calculated and data is presented for Weeks 49-52. Baseline was defined as the average score from the 7 days of eDiary data collected prior to Day 1. Change from Baseline = Post-baseline value minus Baseline value.
Time Frame: Baseline and Weeks 49 to 52
Population: ITT Population
Measure: Median (Full Range); unit: Scores on a scale
Arm/Group | Placebo | Mepolizumab 100 mg SC
Number analyzed (Participants) | 201 | 206
Scores on a scale | -0.90 [-9.11 to 1.19] | -4.48 [-10.00 to 1.62]
Statistical Analysis 1: Comparison: Placebo vs Mepolizumab 100 mg SC; Test type: Other; p = 0.003, Wilcoxon rank-sum test — p-Value was based on Wilcoxon rank-sum test and is adjusted for multiplicity; Difference in Medians = -3.18, 95% CI 2-sided [-4.10 to -2.26] — [estimate comment as in outcome 2, analysis 1]

5. Secondary Outcome: Change From Baseline in Sino-nasal Outcome Test (SNOT)-22 Total Score at Week 52
Description: The SNOT-22 is a 22-item self-reported questionnaire developed to measure symptoms and impacts related to chronic rhinosinusitis. The 22 questions are self-completed by participants based on their recall of their symptoms over the previous 2 weeks using a 6-point rating scale (0 = Not present/no problem; 1 = Very mild problem; 2 = Mild or slight problem; 3 = Moderate problem; 4 = Severe problem; 5 = Problem as "bad as it can be"). Scores for each question are summed to derive the total score. The SNOT-22 total score ranges from 0 to 110, with higher scores representing worse quality of life. Data up to Week 52, including from participants who remained in the study after early discontinuation from IP, were included in analysis. Baseline was defined as Day 1 value. Change from Baseline = Post-baseline value minus Baseline value.
Time Frame: Baseline (Day 1) and Week 52
Population: ITT Population. Only those participants with data available at the specified data point were analyzed.
Measure: Median (Full Range); unit: Scores on a scale
Arm/Group | Placebo | Mepolizumab 100 mg SC
Number analyzed (Participants) | 198 | 205
Scores on a scale | -14.0 [-86 to 38] | -30.0 [-93 to 42]
Statistical Analysis 1: Comparison: Placebo vs Mepolizumab 100 mg SC; Test type: Other; p = 0.003, Wilcoxon rank-sum test — p-Value was based on Wilcoxon rank-sum test and is adjusted for multiplicity; Difference in Medians = -16.49, 95% CI 2-sided [-23.57 to -9.42] — Quantile regression with covariates: treatment, region, Baseline score, Baseline BEC. Par. with nasal surgery prior to Wk 52/withdrew early with no nasal surgery assigned their worst observed score prior to nasal surgery/study withdrawal

6. Secondary Outcome: Percentage of Participants Requiring at Least One Course of Systemic Steroids for Nasal Polyps up to Week 52
Description: The number of courses of systemic steroids received by participants were recorded. For the purpose of this study, a course of systemic corticosteroid separated by less than 7 days was considered as a continuation of the same course. Percentage of participants requiring at least one course of systemic steroids for nasal polyps up to Week 52 is presented. Data up to Week 52, including from participants who remained in the study after early discontinuation from IP, were included in analysis.
Time Frame: Up to Week 52
Population: ITT Population
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Mepolizumab 100 mg SC
Number analyzed (Participants) | 201 | 206
Percentage of participants | 37 | 25
Statistical Analysis 1: Comparison: Placebo vs Mepolizumab 100 mg SC; Test type: Other; p = 0.020, Regression, Logistic — p-Value was based on logistic regression model and is adjusted for multiplicity; Odds Ratio (OR) = 0.58, 95% CI 2-sided [0.36 to 0.92] — Covariates: treatment group, geographic region, number of oral corticosteroids courses for NP in last 12 months(0,1,>1 as ordinal), Baseline total endoscopic score(centrally read),Baseline nasal obstruction VAS score,log(e) Baseline eosinophil count

7. Secondary Outcome: Change From Baseline in the Composite VAS Score (Combining VAS Scores for Nasal Obstruction, Nasal Discharge, Mucus in the Throat and Loss of Smell) During the 4 Weeks Prior to Week 52
Description: Participants rated individual (nasal obstruction, nasal discharge, mucus in the throat, loss of smell, facial pain) and overall symptoms on a visual analog scale using an eDiary. Captured scores ranged between 0 (none) and 100 (as bad as you can imagine), final scores derived from electronically captured scores by dividing by 10. The composite VAS score was calculated as average of individual scores of nasal obstruction, nasal discharge, mucus in the throat and loss of smell and ranged between 0 and 10, with higher scores indicating greater disease severity. Data up to Week 52, including from participants who remained in the study after early discontinuation from IP, were included in analysis. The average of daily scores in 4-weekly intervals were calculated and data is presented for Weeks 49-52. Baseline was defined as the average score from the 7 days of eDiary data collected prior to Day 1. Change from Baseline = Post-baseline value minus Baseline value.
Time Frame: Baseline and Weeks 49 to 52
Population: ITT Population
Measure: Median (Full Range); unit: Scores on a scale
Arm/Group | Placebo | Mepolizumab 100 mg SC
Number analyzed (Participants) | 201 | 206
Scores on a scale | -0.89 [-9.29 to 2.90] | -3.96 [-9.93 to 1.37]
Statistical Analysis 1: Comparison: Placebo vs Mepolizumab 100 mg SC; Test type: Other; p = 0.020, Wilcoxon rank-sum test — p-Value was based on Wilcoxon rank-sum test and is adjusted for multiplicity; Difference in Medians = -2.68, 95% CI 2-sided [-3.44 to -1.91] — [estimate comment as in outcome 2, analysis 1]

8. Secondary Outcome: Change From Baseline in Individual VAS Symptom Score: Loss of Smell During the 4 Weeks Prior to Week 52
Description: Participants rated individual (nasal obstruction, nasal discharge, mucus in the throat, loss of smell, facial pain) and overall symptoms on a visual analog scale using an eDiary. Captured scores ranged between 0 (none) and 100 (as bad as you can imagine), final scores derived from the electronically captured scores by dividing by 10. The final loss of smell VAS score ranged between 0 and 10, with higher scores indicating greater disease severity. Data up to Week 52, including from participants who remained in the study after early discontinuation from IP, were included in analysis. The average of daily scores in 4-weekly intervals were calculated and data is presented for Weeks 49-52. Baseline was defined as the average score from the 7 days of eDiary data collected prior to Day 1. Change from Baseline = Post-baseline value minus Baseline value.
Time Frame: Baseline and Weeks 49 to 52
Population: ITT Population
Measure: Median (Full Range); unit: Scores on a scale
Arm/Group | Placebo | Mepolizumab 100 mg SC
Number analyzed (Participants) | 201 | 206
Scores on a scale | 0.00 [-9.97 to 1.94] | -0.53 [-10.00 to 1.27]
Statistical Analysis 1: Comparison: Placebo vs Mepolizumab 100 mg SC; Test type: Other; p = 0.020, Wilcoxon rank-sum test — p-Value was based on Wilcoxon rank-sum test and is adjusted for multiplicity; Difference in Medians = -0.37, 95% CI 2-sided [-0.65 to -0.08] — [estimate comment as in outcome 2, analysis 1]

ADVERSE EVENTS:
Time Frame: Non-serious adverse events (AEs) and serious AEs were collected from start of study treatment (Day 1) up to Week 52 for treatment period and up to 6 months during no-treatment follow-up period after Week 52 visit
Description: Non-serious AEs and serious AEs were collected for Safety Population which consisted of all randomized participants who took at least one dose of study treatment. Adverse events are presented treatment-wise and period-wise.
Groups:
- Placebo (Treatment Period): Participants were randomized to receive up to 13 SC doses of mepolizumab matching placebo every 4 weeks to Week 52 on top of SoC for nasal polyps which included daily mometasone furorate nasal spray.
- Mepolizumab 100 mg SC (Treatment Period): Participants were randomized to receive up to 13 SC doses of mepolizumab 100 mg/mL every 4 weeks to Week 52 on top of SoC for nasal polyps which included daily mometasone furorate nasal spray.
- Placebo (Follow-up): Participants entered in a 6-month no-treatment follow-up period to assess maintenance of response after cessation of treatment. Participants received mepolizumab matching placebo during treatment period.
- Mepolizumab 100 mg SC (Follow-up): Participants entered in a 6-month no-treatment follow-up period to assess maintenance of response after cessation of treatment. Participants received mepolizumab 100 mg/mL during treatment period.
Arm/Group | Placebo (Treatment Period) | Mepolizumab 100 mg SC (Treatment Period) | Placebo (Follow-up) | Mepolizumab 100 mg SC (Follow-up)
All-Cause Mortality (participants affected / at risk) | 0/201 | 0/206 | 1/65 | 0/69
Serious Adverse Events (participants affected / at risk) | 14/201 | 12/206 | 4/65 | 2/69
Other Adverse Events (participants affected / at risk) | 141/201 | 139/206 | 13/65 | 14/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (Treatment Period) (N=201) | Mepolizumab 100 mg SC (Treatment Period) (N=206) | Placebo (Follow-up) (N=65) | Mepolizumab 100 mg SC (Follow-up) (N=69)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anal polyp (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Benign vulval neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Facial paralysis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Focal segmental glomerulosclerosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastritis erosive (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Migraine with aura (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nephrotic syndrome (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Periorbital cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Uterine polyp (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (Treatment Period) (N=201) | Mepolizumab 100 mg SC (Treatment Period) (N=206) | Placebo (Follow-up) (N=65) | Mepolizumab 100 mg SC (Follow-up) (N=69)
Nasopharyngitis (Infections and infestations) | 46 (64) | 52 (83) | 4 (6) | 6 (8)
Headache (Nervous system disorders) | 44 (141) | 37 (114) | 5 (14) | 5 (8)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 18 (20) | 17 (24) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 22 (29) | 10 (12) | 0 (0) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 14 (16) | 15 (24) | 0 (0) | 0 (0)
Acute sinusitis (Infections and infestations) | 13 (18) | 13 (17) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 10 (11) | 16 (19) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 14 (18) | 12 (20) | 0 (0) | 0 (0)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 16 (28) | 8 (11) | 1 (1) | 3 (3)
Bronchitis (Infections and infestations) | 13 (16) | 10 (10) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 17 (20) | 4 (31) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 13 (15) | 7 (9) | 2 (3) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (6) | 13 (14) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 9 (11) | 8 (11) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 8 (10) | 7 (7) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 10 (12) | 5 (5) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 6 (9) | 7 (12) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 8 (10) | 5 (5) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 5 (5) | 7 (11) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 8 (14) | 4 (5) | 2 (2) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (3) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-02-13): https://cdn.clinicaltrials.gov/large-docs/97/NCT03085797/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-20): https://cdn.clinicaltrials.gov/large-docs/97/NCT03085797/SAP_001.pdf